CLINICAL TRIAL: NCT00761306
Title: A Long-term, Open-label Study Evaluating the Safety and Tolerability of [Vortioxetine] Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: Open-label Safety Extension Study of 5 and 10 mg of Vortioxetine (Lu AA21004) in Long-term Treatment of Major Depressive Disorder in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11492C; 2007-000905-31 (EudraCT Number)
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Long-term; Safety; Open-label
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — 5 or 10 mg/day; tablets; orally
  Other Names: Brintellix

SUMMARY:
The purpose of the study is to evaluate long-term safety and tolerability of Vortioxetine over a period of 52 weeks in patients with Major Depressive Disorder (MDD) having completed 6-week acute treatment in study NCT00839423 / 11492A.

ELIGIBILITY:
Inclusion Criteria:

- Patients who completed 6-week short-term treatment study for Major Depressive Episode (MDE), NCT00839423 / 11492A, followed by a 2-week taper period

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV TR)
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible to participate in present study, NCT00761306 / 11492C, were outpatients, who had completed lead-in study NCT00839423 / 11492A immediately prior to inclusion into present study.
Pre-assignment Details: The study consisted of a 1-week, fixed-dose period with Vortioxetine 10 mg/day, a 51-week flexible dose period with Vortioxetine 5 or 10 mg/day, and a 4-week safety follow up period.
Groups:
- Vortioxetine 5 or 10 mg/Day: tablets; orally
Period: Overall Study
Arm/Group | Vortioxetine 5 or 10 mg/Day
Started | 74
Completed | 54
Not Completed | 20
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 4
Not completed — Protocol Violation | 2
Not completed — Withdrawal of Consent | 3
Not completed — Lost to Follow-up | 1
Not completed — Administrative or Other Reasons | 5

BASELINE CHARACTERISTICS:
Population: Age and Sex: all-patients-treated set (APTS) - all patients who took at least one dose of Vortioxetine in Study NCT00761306 / 11492C; MADRS and HAM-D-24: full-analysis set (FAS) = 74 - all patients in the APTS who had at least one valid Baseline and one valid post-Baseline assessment of the MADRS total score in Study NCT00761306 / 11492C.
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 29
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 10.7 (8.4)
HAM-D-24 [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
  units on a scale | 10.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Time Frame: Up to 52 weeks and a 4-week safety follow-up period
Population: APTS
Measure: Number; unit: participants
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 74
participants
  Patients With AEs | 64
  Patients With SAEs | 1
  Patients With AEs Leading to Withdrawal | 5
  Patients With Baseline Events | 16

2. Primary Outcome: Percentage of Patients Who Withdrew Due to Intolerance to Treatment
Time Frame: Baseline to Week 52
Population: APTS
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 74
percentage of patients | 6.8

3. Secondary Outcome: Change From Baseline in MADRS Total Score After 52 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 55
units on a scale | -4.33 (9.24)

4. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 52 Weeks of Treatment
Description: The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS; OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 59
units on a scale | -3.46 (8.72)

5. Secondary Outcome: Proportion of Responders at Week 52 (Response Defined as a >=50% Decrease in MADRS Total Score)
Time Frame: Week 52
Population: FAS; OC
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 55
percentage of patients | 92.7

6. Secondary Outcome: Proportion of Remitters at Week 52 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 52
Population: FAS; OC
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 5 or 10 mg/Day
Number analyzed (Participants) | 55
percentage of patients | 81.8

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 52-week open label period and 4-week safety follow-up period Other Adverse Events: 52-week open label period
Arm/Group | Vortioxetine 5 or 10 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/74
Other Adverse Events (participants affected / at risk) | 53/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 5 or 10 mg/Day (N=74)
Thyroiditis (Endocrine disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 5 or 10 mg/Day (N=74)
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 5
Gastroenteritis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 17
Weight increased (Investigations) | 14
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. H. Lundbeck A/S follows the Vancouver declaration with respect to authorship.